CLINICAL TRIAL: NCT02346227
Title: Efficiency of AV2 Antiviral Drug in the Treatment of Human Papillomavirus-associated Precancerous Lesions of the Uterine Cervix: a Randomized Clinical Trial in Kinshasa, Democratic Republic of the Congo
Brief Title: Impact of AV2 Antiviral Drug on the Treatment of HPV-associated Lesions of the Uterine Cervix
Acronym: KINVAV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jean-Pierre Van geertruyden (Other)
Collaborators: University of Kinshasa (Other); University Hospital, Antwerp (Other)
Responsible Party: Sponsor-Investigator, Jean-Pierre Van geertruyden, Prof, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UA-IHU- 2012-01
Record Dates: First submitted 2014-11-08; First posted 2015-01-26 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Uterine Cervical Dysplasia; Papillomavirus Infections
Keywords: Human Papillomavirus; Uterine cervix; Infection; Antiviral Drug; Therapeutic use
MeSH Terms: conditions — Uterine Cervical Dysplasia; Papillomavirus Infections; Infections | interventions — lime; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AV2 (Active Comparator): Drug: application of topical spray on the cervix one time (2 puffs) topical application of 100µl AV2 antiviral spray( natural essential oil components in equal volumes diluted 50% in olive oil)
  Interventions: Drug: AV2
- Placebo (Placebo Comparator): Drug: application of topical spray on the cervix one time (2 puffs) topical spray of 100 µl on the cervix.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AV2 — The virucide AV2 consists of a spray. It is a mixture of natural essential oil components (Carvone, Eugenol, Geraniol, Nerolidol) in equal volumes diluted 50% in olive oil (Olea europaea).
  It is administered as a topical spray to the cervix while the subject is in the lithotomic position and fitted with a speculum. The manual spray applicator is positioned inside the anterior of the vagina and two pumps are applied. Each pump delivers 100 microliters of the solution.
  Other Names: Antivirus 2
  Arms: AV2
Drug: Placebo — The placebo consists of 10% lemon (citrus limon) and 10% lime (citrus aurantifolia) in 80% olive oil.
  It is administered as a one time (2 puffs) topical spray of 100 microliters on the cervix.
  Other Names: lemon, lime & olive oil.
  Arms: Placebo

SUMMARY:
1. Introduction Cervical cancer (CC) is a major public health problem in Low-income countries (LICs), particularly in the Democratic Republic of the Congo (DRC), where the estimated number of cases is 3839 per year. (WHO, 2010).

   Persistent infection with Human Papillomavirus (HPV) is recognized as the necessary cause for the development of CC. Thus, CC is a disease that is easily preventable primarily by vaccination against HPV and secondarily through screening and treatment of precancerous lesions of the cervix.

   In LICs, the high incidence of CC is due to both high rates of infection with HPV, a failure to initiate and sustain effective screening programs based on cytology and the non-availability of vaccination against HPV. These situations highlight the need to implement simple and inexpensive screening and treatment methods suitable for LICs. These methods include screening by visual inspection of the cervix after application of acetic acid (VIA) and treatment with a topical antiviral drug (AV2).
2. Aims

   This study aims to:
   * Evaluate the clinical efficacy of AV2 as a treatment for HPV-associated lesions of the uterine cervix;
   * Identify HPV genotypes found in Kinshasa;
   * Determine the cost-effectiveness of an algorithm combining screening by VIA and AV2 and that combining VIA and cryotherapy treatment;
3. Methods After basic training of local health workers on VIA, on collection of cervical samples for HPV testing (quantitative Polymerase Chain reaction, qPCR) and liquid-based cytology (LBC) and on application of AV2, a screening and treatment program will be offered to women aged 25 and older who will give their informed consent.

All women with lesions on VIA will be randomized into one of two groups to receive either treatment by AV2 or placebo.

All women with lesions on VIA will be monitored and reviewed after two months and after six months for repeat tests (VIA and LBC for lesions, qPCR for viral load, conversion and reinfection rates).

DETAILED DESCRIPTION:
CHAPTER 1: INTRODUCTION 1.1. BACKGROUND Cervical cancer (CC) is the third most common cancer in women, and the seventh overall, with an estimated 530 000 new cases per year. More than 85% of the global burden occurs in low-income countries (LICs). It is responsible for 275 000 deaths per year, about 88% of which occurring in LICs. Overall, the mortality: incidence ratio is 52. (Ferlay et al, 2010).

The link between genital high-risk Human papillomavirus (HPV) infections and CC was first demonstrated in the early 1980s by Harold zur Hausen, a German virologist. (Gissmann, L et al, 1983) HPV infection may be transient or persistent. When it persists, HPV induces changes in cells of the cervix, precisely in the transformation zone. These changes constitute the precursor lesions of cervical cancer. These precursor lesions are either called precancerous lesions, dysplasia or cervical intraepithelial neoplasia (CIN). Left untreated, they can progress from mild (CIN1) to moderate (CIN 2) to severe (CIN 3) dysplasia, and then to cancer. It appears that dysplasia is asymptomatic and progresses to cancer over a prolonged period of time, usually 7 to 20 years.

CC is then a potentially preventable and curable cancer. It can be prevented by vaccination against HPV and by screening. The latter involves the detection and treatment of precursors lesions on asymptomatic women.

Several tests can be used for CC screening:

* Cytology (conventional or liquid-based) also called Pap test or Pap smear.
* Visual inspection of the cervix after application of 5% acetic acid or vinegar (VIA).
* HPV-DNA testing. In LIC, the method of screening with low-cost test such as VIA and treating women with positive result with such treatment as cryotherapy in one single visit is known as the "see-and-treat approach". This would minimize loss to follow up, delay in treatment and missed cases.

1.2 ISSUES In HICs, cytology has been introduced as a screening test and reduced markedly the incidence of CC.

In LICs such screening has not been feasible. The high incidence and high mortality for cervical cancer in LIC is due to both high rates of infection with high-risk HPV, a failure to initiate or sustain effective cervical cancer screening programs based on cytology and the non-availability of region-specific HPV vaccine programs.

For that reason, VIA and HPV testing have been recommended for LICs. VIA involves the naked eye inspection of the uterine cervix after application of 3 to 5 % acetic acid. Its sensitivity and negative predictive value are very high, reaching 95% in most of the studies (Sarian, 2005; Sankaranarayanan, 2004).

Only limited data are available on the prevalence and the distribution of HPV variants among women in the general population in DRC. Cytology has been proposed as a screening tool, but it's very opportunistic because there is no organized cervical cancer screening program based on it. On the other hand, most of the Congolese women, living on less than 1 dollar a day can't afford it. Vaccination against HPV infection has not been introduced yet in DRC. It holds promise for the prevention of cervical cancer, yet its impact will not be fully realized until many years after a vaccination program is instituted. To best understand the impact of large-scale vaccination programs, one must first appreciate baseline prevalence of HPV subtypes. Thus, secondary-level prevention i.e. screening is crucial.

Cryotherapy has been proposed as the way to choose for treating cervical precancerous lesions in low-resource settings but it is hampered by major logistic problems (such as availability of carbon dioxide or nitrous oxide); Thus, VIA for screening combined with a simple single treatment with a vaginal spray of AV2 might offer logistical advantages.

1.3 AIMS

Overall Aim:

To contribute to the amelioration of cervical cancer prevention in the Democratic Republic of Congo.

Specific aims:

1. To evaluate the clinical efficacy of the local AV2 antiviral drug in the treatment of HPV-associated cervical lesions.
2. To determine the genotypes of HPV found in the Kinshasa region.
3. To test the impact of HPV screening followed by virucide treatment in a see-and-treat setting on HPV infection and associated cervical lesions.
4. to model the cost-effectiveness of:

   * VIA screening test and virucide treatment algorithm
   * VIA screening test and cryotherapy treatment algorithm 1.4 Hypothesis - The viricidal spray is more effective than placebo in the treatment of HPV-associated cervical precancerous lesions.

CHAPITRE 2: MATERIALS AND METHODS 2.1. Study type and sites: randomized controlled clinical trial. Sites: Centre Hospitalier du Mont-Amba and Centre de santé Lisungi in Kinshasa, D.R. Congo.

Laboratory testing will be performed in a laboratory based in Antwerp, Belgium. 2.2. Population:

* Women aged 25 and over: There is no upper limit in the study population as for the majority of women this will be the first screening contact for HPV and cervical cancer screening. Testing is not performed in women younger than 25 years old as it can be expected that the prevalence of HPV is very high at a younger age and most women will eliminate the virus after some years.
* Sample size and power calculations:

The investigators would like to have enough power in both the HPV-positive group with and without lesions Assuming a HPV clearance rate of 50% in the non-interventional group and 70% in the virucide group at 2 months post-treatment, a minimum sample size of 163 patients (i.e., 124/site) is needed to show with 95% power and 95% certainty a difference between both groups. To allow for up to 10% drop-outs or unevaluable patients, the investigators will recruit at least 190 patients in each arm.

It is supposed that 50 % of those HPV-positive will demonstrate some lesion on VIA, signifying that our secondary randomization on positive lesion will have approximately the same sample size.

The investigators expect 20% of the women to be HPV positive, of whom 10% with and 10% without lesions, indicating that over 1900 ((190*2)/20%) women will have to be enrolled to obtain the required sample size.

As the investigators can screen approximately 50 women per week of whom 70% will be willing and eligible to participate, we expect the study recruitment to last 30 weeks and the time between first recruitment and last patient visit to be 56 weeks.

2.3 Study Design

1. Basic training of doctors working in peripheral health centers where no formal laboratory facilities are available.

   Training will involve VIA and taking cervical swabs for HPV testing and for LBC, not needing any special technical skills; health workers can be trained for these within 1 hour.
2. A local screening program based on VIA will then be offered by these trained doctors to all women aged 25 and over; Samples for qPCR HPV DNA detection, viral load and genotyping and for LBC will also be collected at the same time just before the application of acetic acid. The results of these lab tests will not be available at the moment of randomization and will serve for later analysis.

   The results of the cervical cytology will be reported according to the 2001 Bethesda system terminology.
3. Women showing lesions on VIA will be randomized to one of two groups to receive either AV2 virucide treatment or placebo.

   Women without lesion on VIA will not receive any treatment.
4. All women with lesions will be followed-up and rechecked after two months with VIA, qPCR and LBC.
5. In those testing positive with VIA at the control after 2 months, cryotherapy will be offered as per WHO criteria (Annex 4). It will be performed according to 2011 and 2012 WHO Guidelines and Technical Specifications.
6. In case cervical cancer is detected the patient will be treated according to the local protocol and resources.
7. Six months after the first test, an evaluation including VIA, qPCR and LBC will be performed on all subjects who tested positive at the beginning.
8. Those women with persistent precancerous lesions will be offered appropriate treatment.

Those women without lesion at the beginning but whose HPV test or cytology results will be pathologic will be recalled for appropriate management.

Further treatment will be as per local protocol as at this stage the study ends.

2.4. Statistical analyses Data will be double-entered and cleaned in EpiInfo (version 6.04b, Centers for Diseases Control and Prevention).

Proportions will be compared using the x2 or Fisher's exact tests (when required); Student's t test will be used for continuous variables. A paired t test will be used for within-patient comparisons.

Non-normally distributed variables will be transformed, or nonparametric tests (Wilcoxon or Kruskal-Wallis) will be used.

The log-rank test and the proportional hazard will be estimated (after the Schoenfeld test).

In the case of a proportional hazard regression, all patients will be censored at the time of the last recorded visit.

Stepwise multivariate analyses will be performed, and all possible interactions up to order 2 will be tested.

All reported P values will be 2-sided. For all statistical analyses a P value of ≤ 0.05 will be considered as statistically significant.

All analyses will be performed using the STATA statistical analysis software package (at present version 12; Stata Corp.).

2.5. Ethical issues Regulatory Authorities and Ethical Review Committee This protocol will be submitted for approval by the Institutional ethical committee or Institutional review board (IEC/IRB) of the University of Antwerp and of The Kinshasa School of Public Health and will be registered in an international randomized trial registry before starting.

Patients can be enrolled only after formal approval from the EC

ELIGIBILITY:
Inclusion Criteria:

* Sexually-active women
* Women with intact uterine cervix
* Voluntary written informed consent to participate in the study

Exclusion Criteria:

* Virgin women
* Pregnant or breast-feeding women, and women in the post-partum period
* Subject is already diagnosed with cervical cancer
* Medical history of any severe diseases like hepatitis, renal or liver dysfunction, cardiovascular, gastrointestinal, malignant tumor, or psychiatric disorders etc., which might influence the assessments or conduct of the trial by the discretion of the investigator
* Intake or application of antivirals or other prohibited concomitant medication within 30 days prior to application of AV2®, or patients who plan to take such drugs during the trial
* Known or suspected allergic or adverse response to the investigational product AV2 or its components (olive oil or d-limonene)
* Inability to follow the study protocol

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2015-01; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change of lesions | 2 months
  lesion size" on a scale of 0 - 1 - 2: 0 : for a lesion < 5 mm
  1. : for a lesion 5-15 mm or involving 2 quadrants of the cervix
  2. : for a lesion > 15 mm or involving 3-4 quadrants or endocervically undefined.

SECONDARY OUTCOMES:
absence of HPV DNA | 2 months
  copies/cell
correlation between change of lesions and change in HPV DNA | 2 months
  0 : for a lesion < 5 mm
  1. : for a lesion 5-15 mm or involving 2 quadrants of the cervix
  2. : for a lesion > 15 mm or involving 3-4 quadrants or endocervically undefined. Copies/cell for HPV DNA
Change in HPV viral particle load | 6 months
  copies/cell

OTHER OUTCOMES:
number of patients with adverse effects | 2 months
  Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Yves Jacquemyn, MD PhD, Study Director — University Hospital, Antwerp; Alex Mutombo Baleka, MD, Principal Investigator — University of Kinshasa
Locations (1):
- Centre de Santé Lisungi, Kinshasa, Mont-Ngafula, Democratic Republic of the Congo

REFERENCES:
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Gissmann L, Wolnik L, Ikenberg H, Koldovsky U, Schnurch HG, zur Hausen H. Human papillomavirus types 6 and 11 DNA sequences in genital and laryngeal papillomas and in some cervical cancers. Proc Natl Acad Sci U S A. 1983 Jan;80(2):560-3. doi: 10.1073/pnas.80.2.560. PMID 6300854
- [Background] Sankaranarayanan R, Chatterji R, Shastri SS, Wesley RS, Basu P, Mahe C, Muwonge R, Seigneurin D, Somanathan T, Roy C, Kelkar R, Chinoy R, Dinshaw K, Mandal R, Amin G, Goswami S, Pal S, Patil S, Dhakad N, Frappart L, Fontaniere B. Accuracy of human papillomavirus testing in primary screening of cervical neoplasia: results from a multicenter study in India. Int J Cancer. 2004 Nov 1;112(2):341-7. doi: 10.1002/ijc.20396. PMID 15352050
- [Background] Sarian LO, Derchain SF, Naud P, Roteli-Martins C, Longatto-Filho A, Tatti S, Branca M, Erzen M, Serpa-Hammes L, Matos J, Gontijo R, Braganca JF, Lima TP, Maeda MY, Lorincz A, Dores GB, Costa S, Syrjanen S, Syrjanen K. Evaluation of visual inspection with acetic acid (VIA), Lugol's iodine (VILI), cervical cytology and HPV testing as cervical screening tools in Latin America. This report refers to partial results from the LAMS (Latin AMerican Screening) study. J Med Screen. 2005;12(3):142-9. doi: 10.1258/0969141054855328. PMID 16156945
- [Background] World Health Organization. HPV Summary Report 2010
- [Derived] Baleka Mutombo A, Tozin R, Kanyiki H, Van Geertruyden JP, Jacquemyn Y. Impact of antiviral AV2 in the topical treatment of HPV-associated lesions of the cervix: Results of a phase III randomized placebo-controlled trial. Contemp Clin Trials Commun. 2019 May 16;15:100377. doi: 10.1016/j.conctc.2019.100377. eCollection 2019 Sep. PMID 31193477
- [Derived] Mutombo AB, Tozin R, Simoens C, Lisbeth R, Bogers J, Van Geertruyden JP, Jacquemyn Y. Efficacy of antiviral drug AV2 in the treatment of human papillomavirus-associated precancerous lesions of the uterine cervix: A randomized placebo-controlled clinical trial in Kinshasa, DR Congo. (KINVAV study). Contemp Clin Trials Commun. 2017 Sep 28;8:135-139. doi: 10.1016/j.conctc.2017.09.008. eCollection 2017 Dec. PMID 29696202